CLINICAL TRIAL: NCT04906369
Title: Optimizing Treatment of Metastatic Breast Cancer Through Real-Time Disease Monitoring
Brief Title: Optimizing Treatment of Stage IV Breast Cancer Through Real-Time Disease Monitoring
Status: Suspended | Type: Observational
Why Stopped: lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-001670; NCI-2021-04104 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-05-21; First posted 2021-05-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Patients undergo collection of blood samples at baseline, 2 weeks after the start of treatment, and at the beginning of each new treatment cycle.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples

SUMMARY:
This study evaluates if blood tests can detect changes in disease status during treatment for stage IV breast cancer. Information from this study may help researchers learn more about metastatic breast cancer and how to optimize treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify subtype-specific signatures for breast cancer using genomic positioning of plasma deoxyribonucleic acid (DNA) fragments.

II. To validate changes in circulating tumor-derived DNA (ctDNA) levels as a biomarker for treatment monitoring in patients with metastatic breast cancer.

OUTLINE:

Patients undergo collection of blood samples at baseline, 2 weeks after the start of treatment, and at the beginning of each new treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Stage IV breast cancer undergoing cancer treatment

Exclusion Criteria:

* Stage I-III breast cancer
* Unwilling or unable to give consent
* Patients with a prior or concurrent malignancy, excluding non-melanoma skin cancers and non-invasive cancers whose natural history or treatment does not have the potential to interfere with the assessment of the investigational marker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Mayo Clinic Cancer Center that are undergoing treatment for stage IV breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Identification of patients with high circulating tumor-derived deoxyribonucleic acid (ctDNA) fractions (> 50%) | Up to 1 year
  Will analyze across all three subtypes: Estrogen receptor positive (ER+), human epidermal growth factor receptor 2 positive (HER2+), and triple-negative breast cancer (TNBC). Will perform 30x whole genome sequencing (WGS) and generate subtype-specific pooled nucleosome occupancy maps. By comparing these maps with healthy volunteers, we will identify a set of loci across the genome most informative of cancer contribution in cell-free DNA (cfDNA).
Detection of treatment failure | Up to 1 year
  Defined as progression of disease on imaging studies.

SECONDARY OUTCOMES:
Correlation of shallow whole genome sequencing circulating tumor-derived DNA analysis results with available serologic tumor biomarkers used as a standard in clinical practice | Up to 1 year
  shallow whole genome sequencing circulating tumor-derived DNA analysis results with available serologic tumor biomarkers

OTHER OUTCOMES:
Evaluation of immunity to target antigens and neoantitopes in metastatic breast cancer | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brenda J. Ernst, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States